CLINICAL TRIAL: NCT01982188
Title: Single Incision Suburethral Sling at Time of Robotic Sacrocolpopexy
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Principal Investigator, Atlantic Health System
Other Study IDs: R12-09-001
Record Dates: First submitted 2013-10-31; First posted 2013-11-13 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: single incision sling; cough stress test; MiniArc; UDI-6; UIQ-7; Sandvick Severity Index (SSI)
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single incision sling

SUMMARY:
This study was designed to evaluate urinary function before and one year after single incision sling placement at the time of robotic sacrocolpopexy. The thought is that the more minimally-invasive, single incision sling would provide a similar subjective success rates as those of retropubic and trans-obturator slings.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing single incision sling placement at the time of robotic sacrocolpopexy during the study period

Exclusion Criteria:

* previous surgical treatment for stress urinary incontinence (SUI)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our study population included all women undergoing single incision sling placement at the time of robotic sacrocolpopexy
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cough Stress Test | 12 months post procedure
  Subjects will undergo a cough stress test to evaluate for stress urinary incontinence.

SECONDARY OUTCOMES:
mesh related complications | 12 months post procedure
  possible mesh related complications such as: exposure/erosion, urinary retention, voiding dysfunction, chronic pain and dyspareunia will be collected throughout the study period
Urinary Distress Inventory 6 (UDI-6) | baseline and 12 months postoperatively
  This validated questionnaires will be given to subject to collect subjective data
Urinary Impact Questionnaire (UIQ-7) | baseline and 12 months postoperatively
  this validated questionnaire will be completed by subject to collect subjective data
Sandvick Severity Index Questionnaire | baseline and 12 months postoperatively
  This validated questionnaire will be given to subjects to collect subjective data regarding urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Salamon, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States